CLINICAL TRIAL: NCT04242667
Title: A Randomized Protocol Evaluating Return of Actionable Genetic Research Results to Biobank Participants
Brief Title: Penn Biobank Return of Research Results Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UPCC 08021; 833373 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2020-01-24; First posted 2020-01-27 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Cancer; Cardiovascular Diseases; Hereditary Cancer; Hereditary Cardiac Amyloidosis
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Actionable gene result for cancer risk (Experimental)
  Interventions: Behavioral: e-Health (web-based) disclosure portal; Behavioral: Provider mediated disclosure
- Actionable gene result for cardiovascular disease risk (Experimental)
  Interventions: Behavioral: e-Health (web-based) disclosure portal; Behavioral: Provider mediated disclosure

INTERVENTIONS:
Behavioral: e-Health (web-based) disclosure portal — Patient uses secure web-based portal to access genetic research results
Behavioral: Provider mediated disclosure — Patient has disclosure of genetic research result by a provider (genetic counselor)

SUMMARY:
The overall goal of the proposed research is to assess the feasibility of a randomized study evaluating the non-inferiority of an electronic Health (e-Health) delivery alternative (e.g. private web portal) as compared to return of actionable genetic research results with a genetic counselor.

ELIGIBILITY:
Inclusion Criteria:

1. Consented participant in University of Pennsylvania Biobank who previously submitted a DNA sample for research testing
2. English speaking
3. Aged 18 years or older
4. Agreed to be re-contacted in the future or did not indicate a preference on future contact regarding research results
5. Have an actionable mutation or have been selected as a control participant
6. Have not previously received actionable results of clinical genetic testing

Exclusion Criteria:

1. Deceased assessed by electronic medical record, death index or identified after contact
2. Evidence in the electronic medical record that the subject has already received the same actionable result through clinical genetic testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Completion of surveys | Baseline survey prior to disclosure of results, and then two post-disclosure surveys at 2-7 days and 6 months
  Participant will self-complete surveys to collect psychological and knowledge outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Angela Bradbury, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cocchella G, Phung L, Wood E, Egleston B, Hoffman-Andrews L, Brown S, Ofidis D, Mim R, Griffin H, Fetzer D, Owens A, Domchek S, Pyeritz R, Katona BW, Kallish S, Sirugo G, Weaver J, Nathanson KL, Rader DJ, Bradbury AR. An electronic review of clinical outcomes after return of actionable genetic research results from a health system research biobank. Eur J Med Genet. 2025 Dec;78:105061. doi: 10.1016/j.ejmg.2025.105061. Epub 2025 Nov 13. PMID 41241316